CLINICAL TRIAL: NCT03072654
Title: Thyroidectomy Improves Tracheal Anatomy and Airflow in Patients With Nodular Goiter: A Prospective Cohort Study
Brief Title: Tracheal Anatomy After Thyroidectomy
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Jesper Roed Sorensen, PhD Fellow, University of Southern Denmark
Other Study IDs: S-20130096
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Goiter, Nodular
MeSH Terms: conditions — Goiter, Nodular | interventions — Thyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Thyroidectomy — Remove the nodular goiter on the neck by thyroidectomy (standard procedure)

SUMMARY:
The investigators aimed at investigating the effects of thyroidectomy on tracheal anatomy and airflow in patients with benign nodular goiter, employing a prospective observational study.

Magnetic resonance images of the neck and respiratory flow-volume curves were performed prior to and six months following surgery. Tracheal and thyroid volumes, smallest cross-sectional area of the trachea (SCAT), tracheal narrowing, tracheal deviation and tracheal encirclement by the thyroid were evaluated. Through flow-volume curves respiratory function, including both in- and expiration, was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Reads and write Danish

Exclusion Criteria:

* Suspected or present malignancy
* Neuromuscular disease
* Prior surgery to the neck

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for thyroidectomy for symptomatic benign nodular goiter
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
Changes in tracheal anatomy | 6 months follow-up
  Change in tracheal narrowing (cross sectional area of the trachea at the goiter level compared to cross-sectional area of the trachea at the carina)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brinch FA, Dossing H, Nguyen N, Bonnema SJ, Hegedus L, Godballe C, Sorensen JR. The Impact of Esophageal Compression on Goiter Symptoms before and after Thyroid Surgery. Eur Thyroid J. 2019 Jan;8(1):16-23. doi: 10.1159/000493542. Epub 2018 Oct 17. PMID 30800637